CLINICAL TRIAL: NCT04576676
Title: Environmental Epidemiology of Essential Tremor
Acronym: RULET
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Purdue University (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Yale University (Other)
Responsible Party: Principal Investigator, Elan Louis, Professor and Chairman of Neurology, University of Texas Southwestern Medical Center
Other Study IDs: STU-2020-0563; R01NS094607 (NIH)
Record Dates: First submitted 2020-09-29; First posted 2020-10-06 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Essential Tremor; Parkinson Disease
MeSH Terms: conditions — Essential Tremor; Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 2 vials of veinous blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Essential Tremor: 1. Subjects must be 50 years of age or older.
  2. Subjects must have been diagnosed with Essential Tremor
  3. Subjects must live within 3 hours of UTSW
  Subjects will be screened for eligibility over the phone, and if eligible, will partake in a virtual video conference with a research assistant. Subjects will also travel to the Aston Building at UTSW for a blood draw.
- Parkinson's Disease: 1. Subjects must be 50 years of age or older.
  2. Subjects must have been diagnosed with Parkinson's Disease
  3. Subjects must live within 3 hours of UTSW
  Subjects will be screened for eligibility over the phone, and if eligible, will partake in a virtual video conference with a research assistant. Subjects will also travel to the Aston Building at UTSW for a blood draw.
- Healthy Individuals: 1. Healthy individuals living within 3 hours of UTSW
  2. Subjects must be 50 years of age or older
  3. You are healthy and have not being diagnosed with any neurological disease
  Subjects will be screened for eligibility over the phone, and if eligible, will partake in a virtual video conference with a research assistant. Subjects will also travel to the Aston Building at UTSW for a blood draw.
- Essential Tremor and Parkinson's Disease: 1. Subjects must be 50 years of age or older.
  2. Subjects must have been diagnosed with Essential Tremor
  3. Subjects must have been diagnosed with Parkinson's Disease preceded by at least 3 years of enrollment in study
  4. Subjects must live within 3 hours of UTSW
  Subjects will be screened for eligibility over the phone, and if eligible, will partake in a virtual video conference with a research assistant. Subjects will also travel to the Aston Building at UTSW for a blood draw.

SUMMARY:
This study's research is devoted to studying the causes of tremor, and especially essential tremor (ET), which is the most common type of tremor. Previous studies have revealed a link between harmane [HA], a dietary neurotoxin, and ET; these studies now also suggest a link between this toxin and Parkinson's disease (PD), a related tremor disorder. Yet these links are tentative rather than conclusively established; therefore, in this new patient-based proposal, which incorporates investigations spanning two continents (North America and Europe), utilizes several complementary study designs (prospective cohort, case control), and draws on several types of tissue (blood, brain), the investigator's goal is to nail down the links between HA and ET and to further solidify the emerging links between HA and PD.

DETAILED DESCRIPTION:
This research is devoted to studying the causes of tremor, and especially essential tremor (ET), which is the most common type of tremor. Since 2000, this lab has been investigating whether several environmental neurotoxins are associated with ET. A link between harmane (HA) (1-methyl-9H-pyrido[3,4-b]indole) and ET has been emerging from these studies, which show that blood and brain HA concentration ([HA]) is elevated in ET cases (esp. familial ET) vs. control subjects. HA is a neurotoxin present in the diet (esp. in meat). Administration of HA to laboratory animals produces severe action tremor resembling ET. Yet the link between HA and ET has not been convincingly established. All epidemiological studies have been case-control studies; thus, it is not clear whether high blood [HA] precedes the onset of ET. Aim 1 of this proposal will address this issue. The HA story has also become more complex and multi-dimensional. Thus, the investigators were recently intrigued to find that blood [HA] was higher in Parkinson's disease (PD) cases than controls in New York. HA is structurally similar to MPTP, a neurotoxin closely linked with PD. ET and PD are both tremor disorders; some patients develop both disorders (ET+PD; i.e., they are comorbid for the two conditions). Whether the HA - PD link is reproducible, whether it tracks with the subtype of PD in which tremor rather than bradykinesia/rigidity is the predominant feature, and whether biomarker findings from blood also occur in the target organ of interest (i.e., the brain) in PD is not known. Aim 2 of this proposal will address this myriad of issues. Finally, whether individuals who are comorbid for both ET and PD have the highest blood [HA] is not known. Aim 3 of this proposal will address this issue. To close these gaps in knowledge, in this application, the investigators propose a 5-year study with 3 inter-related aims that draw on several types of human tissue (blood, brain): AIM 1: To nail down the links between HA and ET by studying the association between baseline blood [HA] and the development of incident ET in a cohort study. AIM 2: To further solidify the emerging links between HA and PD by extending our observations to another country (Spain). AIM 3: To assess blood levels of HA in patients who have both ET and PD (ET+PD). This would be the only study heading in this direction - exploring the etiological role of environmental factors, and more specifically toxins, in ET. It would thus complement the many ongoing studies searching for ET genes. The study could lead to the clear identification of the first modifiable risk factor for ET (i.e., dietary HA).This would also be the only study assessing the possible etiological role and tissue concentrations of this toxin, HA, which is structurally similar to MPTP, in patients with PD.

ELIGIBILITY:
Inclusion Criteria:

* Essential Tremor

  * Subjects must be 50 years of age or older.
  * Subjects must have been diagnosed with Essential Tremor
  * Subjects must live within 3 hours of UTSW
* Parkinson's Disease

  * Subjects must be 50 years of age or older.
  * Subjects must have been diagnosed with Parkinson's Disease
  * Subjects must live within 3 hours of UTSW
* Healthy Individuals

  * Healthy individuals living within 3 hours of UTSW
  * Subjects must be 50 years of age or older
  * You are healthy and have not being diagnosed with any neurological disease
* Essential Tremor and Parkinson's Disease

  * Subjects must be 50 years of age or older.
  * Subjects must have been diagnosed with Essential Tremor
  * Subjects must have been diagnosed with Parkinson's Disease preceded by at least 3 years of enrollment in study
  * Subjects must live within 3 hours of UTSW

Exclusion Criteria:

* Healthy Individuals

  * Subjects with medical history of neurological conditions
  * Subjects with family history of neurological condition
  * Subjects with spouse diagnosed with Essential Tremor or Parkinson's Disease
* Essential Tremor

  * Subjects with medical history of another movement disorder such as Parkinson's Disease or dystonia
  * Subjects with head tremor that preceded hand tremor
* Parkinson's Disease

  --Subjects with medical history of Essential Tremor
* Essential Tremor and Parkinson's Disease

  * Criteria that does not meet inclusion

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals above the age of 50, living within a 3 hour driving radius of UT Southwestern.
Sampling Method: Non-Probability Sample
Enrollment: 1497 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2023-07-19 (Actual)

PRIMARY OUTCOMES:
Level of Harmane in Blood | Day 1
  Two vials of veinous blood will be collected from each participant and analyzed for the level of harmane. Specimen collection done at the Aston Care Center and sent to Purdue University for analysis.
Archimedes Spirals | Day 1
  Each participant will draw two spirals with each hand, used to assess the frequency and severity of one's tremor and to confirm their diagnosis.
Video Interview | Day 1
  After a participant has met the eligibility criteria, they participate in a two hour video interview, where a series of questionnaires is administered, as well as a videotaped neurological/movement assessment. Video is reviewed by study's PI and participant's tremor is rated on a fixed, numerical scale from 0.0 to 4.0, where 4.0 indicates a more severe tremor.

SECONDARY OUTCOMES:
Cumulative Illness Rating Scale (CIRS) | Day 1
  CIRS quantifies the burden of disease in elderly patients (comorbidity scale; ranges from 0-42 where 42 indicates highest number and severity of illnesses measured).
Montreal Cognitive Assessment (MoCA) | Day 1
  The MoCA is a cognitive screening test designed to assist Health Professionals in the detection of mild cognitive impairment and Alzheimer's disease. Scores range from 0-30.
Food Frequency Questionnaire | Day 1
  Developed at Harvard University, the Food Frequency Questionnaire (FFQ) is a limited checklist of foods and beverages with a frequency response section for subjects to report how often each item was consumed over a specified period of time.
Meat Questionnaire | Day 1
  Asks participants to indicate how often they eat chicken, beef and pork products, and how well done the meats were cooked.
MDS-Unified Parkinson's Disease Rating Scale | Day 1
  The UPDRS scale refers to Unified Parkinson Disease Rating Scale, and it is a rating tool used to gauge the course of Parkinson's disease in patients. Each of the ratings ranges from 0 to 4. The original UPDRS included only integers, but some use 0.5 increments; however, use of these 0.5 increments has not undergone clinimetric testing or validation. The total score for subscale 3 ranges from 0 to 108, the sum of scores from 27 observations.
Apathy Evaluation Scale (AES) | Day 1
  The Apathy Evaluation Scale (AES) is a method for measuring apathy resulting from brain-related pathology.
Beck's Depression Inventory | Day 1
  The Beck Depression Inventory (BDI, BDI-1A, BDI-II) is a 21-question multiple-choice self-report inventory, one of the most widely used psychometric tests for measuring the severity of depression.
  Like the BDI, the BDI-II also contains 21 questions, each answer being scored on a scale value of 0 to 3. Higher total scores indicate more severe depressive symptoms. The standardized cutoffs used differ from the original:
  0-13: minimal depression 14-19: mild depression 20-28: moderate depression 29-63: severe depression.
Epworth Sleepiness Scale | Day 1
  The ESS is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3), their usual chances of dozing off or falling asleep while engaged in eight different activities. Most people engage in those activities at least occasionally, although not necessarily every day. The ESS score (the sum of 8 item scores, 0-3) can range from 0 to 24. The higher the ESS score, the higher that person's average sleep propensity in daily life (ASP), or their 'daytime sleepiness'.
Hamilton Anxiety Rating Scale (HAM-A) | Day 1
  The HAM-A was one of the first rating scales developed to measure the severity of anxiety symptoms. Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
Patient Health Questionnaire-9 | Day 1
  The Patient Health Questionnaire (PHQ)-9 is the major depressive disorder (MDD) module of the full PHQ. Used to provisionally diagnose depression and grade severity of symptoms in general medical and mental health settings.
Pittsburgh Sleep Quality Index | Day 1
  PSQI was designed to evaluate overall sleep quality. A total score of "5" or greater is indicative of poor sleep quality.
The Snaith-Hamilton Pleasure Scale (SHAPS) | Day 1
  The SHAPS is a 14-item scale that measures anhedonia, the inability to experience pleasure. The items cover the domains of: social interaction, food and drink, sensory experience, and interest/pastimes. A score of 2 or less constitutes a "normal" score, while an "abnormal" score is defined as 3 or more.
Tremor Disability Questionnaire | Day 1
  Assesses a valid index of tremor-induced disability
Tremor Embarrassment Assessment (TEA) | Day 1
  TEA is a tool to quantitatively assess the level of embarrassment experienced due to one's tremor.

CONTACTS AND LOCATIONS:
Overall Officials: Nora C Hernandez, M.D., Study Director — UTSW Medical Center; Allison Powell, BA, Study Director — UTSW Medical Center
Locations (1):
- University of Texas Southwestern, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
We are committed to making the resources of this study widely available not only to scientists studying ET but to those studying other neurological and neurodegenerative diseases as well, and especially to those who are studying PD. Thus, sharing data generated by this project is an important part of our proposed activities and will be carried out in a number of different ways. Our Data Sharing plan will adhere to the general principles outlined in the NIH Data Sharing Policy and Implementation Guidance.
  The aims of the present proposal not only include clinical data but also data from measurement of harmane in blood and brain tissue samples. Data/tissue will be shared for all study participants that have consented to data sharing. Participants who did not give consent for data sharing will be excluded.
Time Frame: Data will become available after the recruitment is complete and the biological samples have been analyzed.
Access Criteria: The results and conclusions of our analysis will be shared at global scientific meetings and in the scientific literature (during publication in peer-reviewed journals). An additional mechanism of sharing data will be in the form of supplements to the additional data, which, for most journals, is on-line.
  The data will be entered into SPSS data files. Original data files for individual runs will be shared with colleagues who possess the means and knowledge to utilize them, under collaborative agreement. To strengthen data confidentiality and safeguard the privacy of study participants, we will make data available to approved researchers under a data-sharing agreement that provides for (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology and (3) a commitment to destroying or returning the data after analyses are completed.

REFERENCES:
- [Background] Louis ED. Clinical practice. Essential tremor. N Engl J Med. 2001 Sep 20;345(12):887-91. doi: 10.1056/NEJMcp010928. No abstract available. PMID 11565522
- [Background] Louis ED, Applegate LM, Factor-Litvak P, Parides MK, Andrews L. Essential tremor: occupational exposures to manganese and organic solvents. Neurology. 2004 Dec 14;63(11):2162-4. doi: 10.1212/01.wnl.0000145600.91491.f2. PMID 15596771
- [Background] Louis ED, Benito-Leon J, Moreno-Garcia S, Vega S, Romero JP, Bermejo-Pareja F, Gerbin M, Viner AS, Factor-Litvak P, Jiang W, Zheng W. Blood harmane (1-methyl-9H-pyrido[3,4-b]indole) concentration in essential tremor cases in Spain. Neurotoxicology. 2013 Jan;34:264-8. doi: 10.1016/j.neuro.2012.09.004. Epub 2012 Sep 12. PMID 22981972
- [Background] Louis ED, Zheng W, Applegate L, Shi L, Factor-Litvak P. Blood harmane concentrations and dietary protein consumption in essential tremor. Neurology. 2005 Aug 9;65(3):391-6. doi: 10.1212/01.wnl.0000172352.88359.2d. PMID 16087903
- [Background] Bhalsing KS, Saini J, Pal PK. Understanding the pathophysiology of essential tremor through advanced neuroimaging: a review. J Neurol Sci. 2013 Dec 15;335(1-2):9-13. doi: 10.1016/j.jns.2013.09.003. Epub 2013 Sep 10. PMID 24060292
- [Background] Benito-Leon J, Louis ED, Bermejo-Pareja F; Neurological Disorders in Central Spain Study Group. Risk of incident Parkinson's disease and parkinsonism in essential tremor: a population based study. J Neurol Neurosurg Psychiatry. 2009 Apr;80(4):423-5. doi: 10.1136/jnnp.2008.147223. PMID 19289477
- [Background] Louis ED, Ferreira JJ. How common is the most common adult movement disorder? Update on the worldwide prevalence of essential tremor. Mov Disord. 2010 Apr 15;25(5):534-41. doi: 10.1002/mds.22838. PMID 20175185
- [Background] Bain PG, Findley LJ, Thompson PD, Gresty MA, Rothwell JC, Harding AE, Marsden CD. A study of hereditary essential tremor. Brain. 1994 Aug;117 ( Pt 4):805-24. doi: 10.1093/brain/117.4.805. PMID 7922467
- [Background] Louis ED, Benito-Leon J, Ottman R, Bermejo-Pareja F; Neurological Disorders in Central Spain (NEDICES) Study Group. A population-based study of mortality in essential tremor. Neurology. 2007 Nov 20;69(21):1982-9. doi: 10.1212/01.wnl.0000279339.87987.d7. PMID 18025392
- [Background] Fekete R, Jankovic J. Revisiting the relationship between essential tremor and Parkinson's disease. Mov Disord. 2011 Feb 15;26(3):391-8. doi: 10.1002/mds.23512. PMID 21462256
- [Background] MARSHALL J. Observations on essential tremor. J Neurol Neurosurg Psychiatry. 1962 May;25(2):122-5. doi: 10.1136/jnnp.25.2.122. No abstract available. PMID 14470250
- [Background] Louis ED, Vonsattel JP, Honig LS, Lawton A, Moskowitz C, Ford B, Frucht S. Essential tremor associated with pathologic changes in the cerebellum. Arch Neurol. 2006 Aug;63(8):1189-93. doi: 10.1001/archneur.63.8.1189. PMID 16908751
- [Background] Moncrieff J. Determination of pharmacological levels of harmane, harmine and harmaline in mammalian brain tissue, cerebrospinal fluid and plasma by high-performance liquid chromatography with fluorimetric detection. J Chromatogr. 1989 Nov 24;496(2):269-78. doi: 10.1016/s0378-4347(00)82576-1. PMID 2613832
- [Background] Skog K, Solyakov A, Arvidsson P, Jagerstad M. Analysis of nonpolar heterocyclic amines in cooked foods and meat extracts using gas chromatography-mass spectrometry. J Chromatogr A. 1998 Apr 17;803(1-2):227-33. doi: 10.1016/s0021-9673(97)01266-1. PMID 9604333
- [Background] Gironell A, Kulisevsky J, Barbanoj M, Lopez-Villegas D, Hernandez G, Pascual-Sedano B. A randomized placebo-controlled comparative trial of gabapentin and propranolol in essential tremor. Arch Neurol. 1999 Apr;56(4):475-80. doi: 10.1001/archneur.56.4.475. PMID 10199338
- [Background] Benito-Leon J, Louis ED, Bermejo-Pareja F; Neurological Disorders in Central Spain (NEDICES) Study Group. Population-based case-control study of cognitive function in essential tremor. Neurology. 2006 Jan 10;66(1):69-74. doi: 10.1212/01.wnl.0000192393.05850.ec. PMID 16401849

DOCUMENTS (1):
  • Informed Consent Form (2022-08-05): https://cdn.clinicaltrials.gov/large-docs/76/NCT04576676/ICF_000.pdf